CLINICAL TRIAL: NCT03051685
Title: Bioavailability of DFN-15 at 3 Different Doses vs. Comparator and to Determine Dose-proportionality of DFN-15 in Fasting Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: DFN-15-CD-003
Record Dates: First submitted 2017-02-07; First posted 2017-02-14 (Actual); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- DFN-15 Dose 1 (Experimental)
  Interventions: Drug: DFN-15 Dose 1
- DFN-15 Dose 2 (Experimental)
  Interventions: Drug: DFN-15 Dose 2
- DFN-15 Dose 3 (Experimental)
  Interventions: Drug: DFN-15 Dose 3
- Active Comparator (Active Comparator)
  Interventions: Drug: Active Comparator

INTERVENTIONS:
Drug: DFN-15 Dose 1
  Arms: DFN-15 Dose 1
Drug: DFN-15 Dose 2
  Arms: DFN-15 Dose 2
Drug: DFN-15 Dose 3
  Arms: DFN-15 Dose 3
Drug: Active Comparator
  Arms: Active Comparator

SUMMARY:
Crossover study to compare the BA of DFN-15 at 3 different doses versus the comparator to determine dose-proportionality of DFN-15 in healthy volunteers under fasting conditions

ELIGIBILITY:
Inclusion Criteria:

Subjects were male or female, at least 18 years of age but not older than 45 years of age. The main inclusion criteria were:

1. non- or ex-smokers
2. body mass index (BMI) ≥18.50 kg/m2 and <30.00 kg/m2
3. no clinically significant abnormality found in the 12-lead ECG performed at study entry
4. negative pregnancy test for female subjects
5. healthy according to medical history, complete physical examination (including vital signs) and laboratory tests (general biochemistry, hematology, urinalysis, and coagulation)
6. Fecal occult blood determination negative at screening

Exclusion Criteria:

1. Females who were pregnant or were lactating
2. Patients who had a history of allergic reactions to non-steroidal anti-inflammatory drugs (NSAIDs), including patients in whom aspirin or other NSAIDs induce the syndrome of asthma, rhinitis, nasal polyps or Samter's triad
3. Presence of significant gastrointestinal, liver or kidney disease, or any other conditions known to interfere with the absorption, distribution, metabolism or excretion of drugs or known to potentiate or predispose to undesired effects
4. History of significant gastrointestinal, liver or kidney disease that may affect drug bioavailability
5. Presence of significant cardiovascular, pulmonary, hematologic, neurological, psychiatric, endocrine, immunologic or dermatologic disease
6. Suicidal tendency, history of or disposition to seizures, state of confusion, clinically relevant psychiatric diseases, neurological impairment or cognitive dysfunction that, in the opinion of the investigator, would compromise validity of informed consent, study participation and compliance or data collection
7. Presence of out-of-range cardiac intervals and/ or morphological changes suggestive of arrhythmias or ischaemic heart disease on the screening electrocardiogram (ECG) or other clinically significant ECG abnormalities
8. History or current hypertension, bleeding disorders, ischaemic heart disease, stroke and/or cerebrovascular disease or renal disease
9. History of asthma, urticaria, or allergic-type reactions after taking acetylsalicylic acid (ASA) or other NSAIDs
10. Presence or history of gastric, duodenal or peptic ulcer or gastrointestinal bleeding
11. Use of ASA or NSAIDs, or any product containing ASA or NSAIDs, in the previous 7 days before day 1 of this study
12. Known presence of rare hereditary problems of galactose and /or lactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption
13. Maintenance therapy with any drug or significant history of drug dependency (including marijuana and medical marijuana) or alcohol abuse (> 3 units of alcohol per day, intake of excessive alcohol, acute or chronic) within 1 year
14. Any clinically significant illness in the previous 28 days before day 1 of this study
15. Any history of tuberculosis and/or prophylaxis for tuberculosis
16. Positive urine screening of alcohol and/or drugs of abuse
17. Positive results to HIV Ag/Ab Combo, Hepatitis B surface Antigen (HBsAG (B)) or anti Hepatitis C Virus (HCV (C)) tests
18. Females who were pregnant according to a positive pregnancy test
19. Volunteers who took an investigational product (in another clinical trial) in the previous 28 days before day 1 of this study or who had already participated in this clinical study
20. Volunteers who donated plasma in the previous 14 days before day 1 of this study
21. Donation of 500 mL or more of blood (American Red Cross, clinical studies, etc.) in the previous 56 days before day 1 of this study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2015-07-20 (Actual); Primary Completion 2015-08-14 (Actual); Study Completion 2015-11-10 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic (PK) parameters of DFN-15 | Up to 72 hours
  DFN-15 maximum Plasma Concentration (Cmax)
Pharmacokinetic (PK) parameters of DFN-15 | 15 minutes
  Area under the curve (AUC) 0-15 min
Pharmacokinetic (PK) parameters of DFN-15 | 30 minutes
  Area under the curve (AUC) 0-30
Pharmacokinetic (PK) parameters of DFN-15 | 1 hour
  Area under the curve (AUC) 0-1 hour
Pharmacokinetic (PK) parameters of DFN-15 | 2 hours
  Area under the curve (AUC) 0-2 hours
Pharmacokinetic (PK) parameters of DFN-15 | Up to 72 hours
  Area under the curve (AUC) 0-T
Pharmacokinetic (PK) parameters of DFN-15 | Up to 72 hours
  Area under the curve (AUC) 0-RefTmax
Pharmacokinetic (PK) parameters of DFN-15 | Up to 72 hours
  Area under the curve (AUC) 0-∞

CONTACTS AND LOCATIONS:
Locations (1):
- Site 1, Fargo, North Dakota, United States

REFERENCES:
- [Result] Pal A, Shenoy S, Gautam A, Munjal S, Niu J, Gopalakrishnan M, Gobburru J. Pharmacokinetics of DFN-15, a Novel Oral Solution of Celecoxib, Versus Celecoxib 400-mg Capsules: A Randomized Crossover Study in Fasting Healthy Volunteers. Clin Drug Investig. 2017 Oct;37(10):937-946. doi: 10.1007/s40261-017-0548-6. PMID 28748412